CLINICAL TRIAL: NCT01006733
Title: Genetics Informatics Trial (GIFT) of Warfarin to Prevent Deep Venous Thrombosis (DVT)
Brief Title: Genetics Informatics Trial (GIFT) of Warfarin to Prevent DVT
Acronym: GIFT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); Hospital for Special Surgery, New York (Other); Intermountain Health Care, Inc. (Other); University of Utah (Other); Rush University Medical Center (Other); University of Texas Southwestern Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Prevention
Other Study IDs: HL097036-01; R01HL097036 (NIH)
Record Dates: First submitted 2009-10-30; First posted 2009-11-03 (Estimated); Last update posted 2016-12-29 (Estimated); Status verified 2016-12

CONDITIONS: Thromboembolism
Keywords: pharmacogenetics; arthroplasty; VKORC1; thromboembolism; warfarin
MeSH Terms: conditions — Thromboembolism; Vitamin K-Dependent Clotting Factors, Combined Deficiency Of, Type 2 | interventions — Pharmacogenomic Testing

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Target INR 1.8 and Pharmacogenetic (Experimental): The target International Normalized Ratio (INR) is 1.8. Warfarin initiation is via Pharmacogenetic dosing.
  Interventions: Genetic: Pharmacogenetic; Drug: Target INR 1.8
- Target INR 2.5 and Pharmacogenetic (Experimental): The target INR is 2.5. Warfarin initiation is via Pharmacogenetic dosing.
  Interventions: Genetic: Pharmacogenetic
- Target INR 1.8 and Clinical (Experimental): The target INR is 1.8. Warfarin initiation is via clinical dosing.
  Interventions: Drug: Target INR 1.8
- Target INR 2.5 and Clinical (No Intervention): The target INR is 2.5. Warfarin initiation is via clinical dosing.

INTERVENTIONS:
Genetic: Pharmacogenetic — The pharmacogenetic arm estimates therapeutic warfarin dose using cytochrome P 450 2C9 (CYP2C9), vitamin K epoxide reductase complex subunit 1 (VKORC1), and cytochrome P 450 4F2 (CYP4F2) genotype and clinical information. The clinical arm estimates warfarin dose from clinical information alone.
  Arms: Target INR 1.8 and Pharmacogenetic; Target INR 2.5 and Pharmacogenetic
Drug: Target INR 1.8 — We will randomize patients to a target International Normalized Ratio (INR) of 2.5 or 1.8.
  Arms: Target INR 1.8 and Clinical; Target INR 1.8 and Pharmacogenetic

SUMMARY:
Blood clots contribute to the death of at least 100,000 Americans each year. Because many of these deaths occur suddenly where treatment is impossible, the best treatment is prevention. With this grant, researchers in Missouri, New York, Utah, Illinois, and Texas are developing strategies to improve the safety and effectiveness of clot prevention by customizing a popular blood thinner (warfarin) to each person's genetic and clinical profile. They hypothesize that the use of genetics to guide warfarin therapy will reduce the risk of venous thromboembolism (VTE) postoperatively. They further hypothesize that using a target international normalized ratio (INR) of 1.8 is non-inferior to using a target INR of 2.5 in VTE prevention.

DETAILED DESCRIPTION:
The overall objective of the Genetics-InFormatics Trial (GIFT) of Warfarin to Prevent DVT is to elucidate novel strategies to improve the safety and effectiveness of warfarin therapy. With this study we directly respond to Health and Human Services (HHS) priorities to advance the field of personalized medicine and to prevent venous thromboembolic (VTE) disease. In 2007, the Honorable Mike Leavitt, Secretary of HHS, announced the Personalized Health Care Initiative and wrote that a key goal was, "… to use our personal genetic information to tailor treatments more effectively to each patient."(1) Recently, President Obama and Francis Collins (Director of the NIH) have made precision medicine a national priority.(2) Previously, the Acting Surgeon General issued a Call to Action to reduce the number of cases of VTE in the United States.(3) To facilitate precision dosing strategies for VTE prevention, we have made publically available a non-profit, web application, www.WarfarinDosing.org. A public version of www.WarfarinDosing.org estimates warfarin doses for the initial 5 days of warfarin therapy. The version being evaluated in GIFT provides doses for the initial 11 days of warfarin therapy.

Aim 1: To determine how pharmacogenetic-based warfarin therapy affects the safety and effectiveness of warfarin therapy. The intensity of anticoagulant therapy is measured by the International Normalized Ratio (INR). During initiation, the INR often falls outside the therapeutic range. INRs that are too low predispose patients to VTE while supratherapeutic INR values increase risk of bleeding.(4, 5) Previously, the FDA approved the label change of warfarin/Coumadin™ to recommend considering lower initial doses in patients known to have certain polymorphisms in genes affecting warfarin metabolism and sensitivity.(6) However, whether this strategy improves the safety and effectiveness of warfarin therapy in general is unknown. In particular, how this strategy affects subgroups with and without the genetic variants of interest is also unknown.

Hypothesis 1: Pharmacogenetic therapy decreases the composite risk of a non-fatal VTE, non-fatal major hemorrhage, death, or INR ≥ 4.0 in all patients, and/or in the subgroup of patients whose pharmacogenetic and clinical predicted therapeutic maintenance doses differ by > 1.0 mg/day. Based on our meta-analysis of prior trials(7), we anticipate 80% power to simultaneously detect a 32% relative risk reduction in the composite outcome for

Aim 1 (as measured by a chi-square test). In the clinical arm, based on preliminary data, we anticipate that the rate of the composite outcome will be 15.7% in the clinical arm and 10.7% in the pharmacogenetic arm. We obtained these estimates because they average a rate of 13.2%, which is the rate of the composite outcome for Aim 1 observed from the initial 775 GIFT participants. The power was calculated using a two-sided alpha of 0.05 for a test of proportions, a drop-out rate of 2%, and a partitioned (two-sided) alpha with 0.044 allocated to the whole population and 0.01 to the high-risk subgroup. Because of correlation between these two subgroups, using these alphas preserves an overall type 1 error rate of 0.05.

Aim 2: To determine whether warfarin therapy with a target INR of 1.8 is non-inferior to therapy with a target INR of 2.5 at preventing VTE or death in orthopedic patients. One randomized trial (PREVENT) found that a target INR value of 1.5-2.0 prevented 64% of VTE recurrence.(8) Although that trial excluded orthopedic patients, such an approach has been endorsed by the American Academy of Orthopedic Surgeons (AAOS). On page 15 of the 2007 AAOS guidelines (9) they offer the following recommendation for VTE prophylaxis around the time of joint replacement: "Warfarin, with an INR goal of ≤ 2.0, starting either the night before or the night after surgery, for 2-6 weeks." However, the AAOS grade the overall evidence for VTE prophylaxis in this population as low (level III). The AAOS guidelines conflict with the prior American College of Chest Physician (ACCP) guidelines,(10) which recommend, as one of their (Grade 1A) options (page 338 S), using an "…adjusted-dose vitamin K antagonist (INR target, 2.5; range 2.0 to 3.0)." Because lower target INR values may reduce the risk of hemorrhage and simplify warfarin management(8) we propose to test the following:

Hypothesis 2: For prevention of non-fatal VTE or death, a target INR of 1.8 will be non-inferior to a higher target INR (2.5). Using a non-inferiority margin of 3% absolute risk reduction in non-fatal VTE or death and an estimated composite rate of 5.56% (based on preliminary GIFT data), we will have 83% power to detect the non-inferiority of a target INR of 1.8 in 1600 patients.

ELIGIBILITY:
Inclusion Criteria:

* 65 years of age or older
* must anticipate taking warfarin for at least 4 weeks for VTE prophylaxis after hip or knee arthroplasty
* must be able to give written, informed consent
* must have venous access
* must not be institutionalized, incarcerated at the time of enrollment (nursing home okay)
* must have life expectancy > 6 months
* must have plans to have regular INR monitoring
* willing/able to follow-up in 3-7 weeks with a Doppler Ultrasound

Exclusion Criteria:

* Baseline INR > 1.35
* knowledge of CYP2C9, VKORC1, or CYP4F2 genotype
* knowledge of warfarin dose requirements from prior warfarin therapy
* absolute contraindication or allergy to warfarin therapy (e.g. pregnancy)
* receiving or planning to receive any anticoagulant besides warfarin (if low molecular weight heparin (LMWH) or subcutaneous heparin is deemed necessary by the clinician after enrollment, such patients will be allowed to remain in the study)
* unlikely to be compliant (e.g. due to history of non-compliance, or alcoholism)
* known thrombophilia, bleeding disorder, or history of serious bleed in the past 2 years (unless caused by trauma)
* personal history of venous thromboembolism

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 1598 (Actual)
Dates: Start 2011-03; Primary Completion 2016-10 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
For Aim 1: The composite outcome of: non-fatal venous thromboembolism (VTE), non-fatal major hemorrhage, INR>=4.0, and death. | 30-days, except that VTE may be detected up to day 60
For Aim 2: The composite outcome of: non-fatal venous thromboembolism (VTE) and death. | 30-days for death; 60 days for VTE

SECONDARY OUTCOMES:
Percent Time in Therapeutic INR Range | 4-28 days
  We also we report INR Variability using the method of Lind et al. (2012 Thrombosis research).
Composite Outcomes | 30 days for death; 60 days for VTE, major bleed, INR >=4.0.
  We will compare the two arms in Aim 2 using the same composite outcome from Aim 1: VTE, major hemorrhage, death, or INR >= 4.0.
Ranked Outcomes | 4-28 days for PTTR (INR variability); 30 days for death; 60 days for VTE.
  Outcomes will be ranked using the following tiers in hierarchical order, from worst to best: (1) death; (2) PE; (3) Major bleed; (4) symptomatic DVT; (5) INR >= 4 with minor bleed; (6) asymptomatic DVT; (7) INR >= 4 (w/out major/minor bleed); (8) PTTR.
  Events that happen earliest receive the lowest (worst) score. For PTTR, lower time in the target INR range is worse. This approach, similar to that used in the RELAX trial (Redfield et al. 2013) weighs outcomes according to their clinical relevance. Ranks will be compared using a standard non-parametric test (Mann-Whitney 1947) to determine if one arm improves outcomes.
Time to first laboratory event (INR > 1.5 + Target INR) | Maximum of 90 days; median time to last INR is 28 days

CONTACTS AND LOCATIONS:
Overall Officials: Brian F Gage, MD, MSc, Principal Investigator — Washington University School of Medicine
Locations (6):
- United States (6):
  - Rush University Medical Center, Chicago, Illinois
  - Washington University in St. Louis, School of Medicine, St Louis, Missouri
  - Hospital for Special Surgery, Weill-Cornell, New York, New York
  - University of Texas Southwestern, Dallas, Texas
  - University of Utah, Salt Lake City, Utah
  - Intermountain Medical Center, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: Yes
GIFT plans to share anonymous IPD with other researchers via BioLINCC in March 2018.

REFERENCES:
- [Background] Lenzini P, Wadelius M, Kimmel S, Anderson JL, Jorgensen AL, Pirmohamed M, Caldwell MD, Limdi N, Burmester JK, Dowd MB, Angchaisuksiri P, Bass AR, Chen J, Eriksson N, Rane A, Lindh JD, Carlquist JF, Horne BD, Grice G, Milligan PE, Eby C, Shin J, Kim H, Kurnik D, Stein CM, McMillin G, Pendleton RC, Berg RL, Deloukas P, Gage BF. Integration of genetic, clinical, and INR data to refine warfarin dosing. Clin Pharmacol Ther. 2010 May;87(5):572-8. doi: 10.1038/clpt.2010.13. Epub 2010 Apr 7. PMID 20375999
- [Background] Ferder NS, Eby CS, Deych E, Harris JK, Ridker PM, Milligan PE, Goldhaber SZ, King CR, Giri T, McLeod HL, Glynn RJ, Gage BF. Ability of VKORC1 and CYP2C9 to predict therapeutic warfarin dose during the initial weeks of therapy. J Thromb Haemost. 2010 Jan;8(1):95-100. doi: 10.1111/j.1538-7836.2009.03677.x. Epub 2009 Oct 30. PMID 19874474
- [Background] King CR, Deych E, Milligan P, Eby C, Lenzini P, Grice G, Porche-Sorbet RM, Ridker PM, Gage BF. Gamma-glutamyl carboxylase and its influence on warfarin dose. Thromb Haemost. 2010 Oct;104(4):750-4. doi: 10.1160/TH09-11-0763. Epub 2010 Aug 5. PMID 20694283
- [Background] Finkelman BS, Gage BF, Johnson JA, Brensinger CM, Kimmel SE. Genetic warfarin dosing: tables versus algorithms. J Am Coll Cardiol. 2011 Feb 1;57(5):612-8. doi: 10.1016/j.jacc.2010.08.643. PMID 21272753
- [Background] Johnson JA, Gong L, Whirl-Carrillo M, Gage BF, Scott SA, Stein CM, Anderson JL, Kimmel SE, Lee MT, Pirmohamed M, Wadelius M, Klein TE, Altman RB; Clinical Pharmacogenetics Implementation Consortium. Clinical Pharmacogenetics Implementation Consortium Guidelines for CYP2C9 and VKORC1 genotypes and warfarin dosing. Clin Pharmacol Ther. 2011 Oct;90(4):625-9. doi: 10.1038/clpt.2011.185. Epub 2011 Sep 7. PMID 21900891
- [Background] Horne BD, Lenzini PA, Wadelius M, Jorgensen AL, Kimmel SE, Ridker PM, Eriksson N, Anderson JL, Pirmohamed M, Limdi NA, Pendleton RC, McMillin GA, Burmester JK, Kurnik D, Stein CM, Caldwell MD, Eby CS, Rane A, Lindh JD, Shin JG, Kim HS, Angchaisuksiri P, Glynn RJ, Kronquist KE, Carlquist JF, Grice GR, Barrack RL, Li J, Gage BF. Pharmacogenetic warfarin dose refinements remain significantly influenced by genetic factors after one week of therapy. Thromb Haemost. 2012 Feb;107(2):232-40. doi: 10.1160/TH11-06-0388. Epub 2011 Dec 21. PMID 22186998
- [Background] Do EJ, Lenzini P, Eby CS, Bass AR, McMillin GA, Stevens SM, Woller SC, Pendleton RC, Anderson JL, Proctor P, Nunley RM, Davila-Roman V, Gage BF. Genetics informatics trial (GIFT) of warfarin to prevent deep vein thrombosis (DVT): rationale and study design. Pharmacogenomics J. 2012 Oct;12(5):417-24. doi: 10.1038/tpj.2011.18. Epub 2011 May 24. PMID 21606949
- [Background] Kawai VK, Cunningham A, Vear SI, Van Driest SL, Oginni A, Xu H, Jiang M, Li C, Denny JC, Shaffer C, Bowton E, Gage BF, Ray WA, Roden DM, Stein CM. Genotype and risk of major bleeding during warfarin treatment. Pharmacogenomics. 2014 Dec;15(16):1973-83. doi: 10.2217/pgs.14.153. PMID 25521356
- [Background] Bass AR, Rodriguez T, Hyun G, Santiago FG, Kim JI, Woller SC, Gage BF. Myocardial ischaemia after hip and knee arthroplasty: incidence and risk factors. Int Orthop. 2015 Oct;39(10):2011-6. doi: 10.1007/s00264-015-2853-0. Epub 2015 Jul 9. PMID 26156715
- [Background] Hyun G, Li J, Bass AR, Mohapatra A, Woller SC, Lin H, Eby C, McMillin GA, Gage BF. Use of signals and systems engineering to improve the safety of warfarin initiation. J Thromb Thrombolysis. 2016 Nov;42(4):529-33. doi: 10.1007/s11239-016-1402-z. PMID 27443162
- [Derived] Gage BF, Bass AR, Lin H, Woller SC, Stevens SM, Al-Hammadi N, Anderson JL, Li J, Rodriguez T Jr, Miller JP, McMillin GA, Pendleton RC, Jaffer AK, King CR, Whipple B, Porche-Sorbet R, Napoli L, Merritt K, Thompson AM, Hyun G, Hollomon W, Barrack RL, Nunley RM, Moskowitz G, Davila-Roman V, Eby CS. Effect of Low-Intensity vs Standard-Intensity Warfarin Prophylaxis on Venous Thromboembolism or Death Among Patients Undergoing Hip or Knee Arthroplasty: A Randomized Clinical Trial. JAMA. 2019 Sep 3;322(9):834-842. doi: 10.1001/jama.2019.12085. PMID 31479138
- [Derived] Gage BF, Bass AR, Lin H, Woller SC, Stevens SM, Al-Hammadi N, Li J, Rodriguez T Jr, Miller JP, McMillin GA, Pendleton RC, Jaffer AK, King CR, Whipple BD, Porche-Sorbet R, Napoli L, Merritt K, Thompson AM, Hyun G, Anderson JL, Hollomon W, Barrack RL, Nunley RM, Moskowitz G, Davila-Roman V, Eby CS. Effect of Genotype-Guided Warfarin Dosing on Clinical Events and Anticoagulation Control Among Patients Undergoing Hip or Knee Arthroplasty: The GIFT Randomized Clinical Trial. JAMA. 2017 Sep 26;318(12):1115-1124. doi: 10.1001/jama.2017.11469. PMID 28973620
- See also: pharmacogenetic and clinical warfarin dosing algorithms for trial — http://www.warfarindosing.org